CLINICAL TRIAL: NCT01833117
Title: A Randomized, Observer-Masked, Efficacy and Safety Study of FID 119515A in Dry Eye
Brief Title: Efficacy and Safety Study of FID 119515A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-12-021
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2014-04

CONDITIONS: Dry Eye
Keywords: Dry eye; Tear film; Tear break-up time; Ocular surface; Eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 119515A (Experimental): FID 119515A, 1 drop instilled in the study eye, single dose
  Interventions: Other: FID 119515A
- Blink (Active Comparator): Blink® Tears, 1 drop instilled in the study eye, single dose
  Interventions: Other: Blink® Tears

INTERVENTIONS:
Other: FID 119515A — topical ocular drops
  Arms: FID 119515A
Other: Blink® Tears — topical ocular drops
  Arms: Blink

SUMMARY:
The purpose of this study was to compare the effect of FID 119515A to Blink® Tears on the integrity of tear film in adults with a history of dry eye in both eyes.

DETAILED DESCRIPTION:
Subjects who met the enrollment criteria were randomized in a 2:1 manner to receive treatment with FID 119515A or Blink® Tears respectively for this 1-day, single-dose study.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* Best corrected visual acuity (BCVA) of 55 or greater in each eye as measured by an ETDRS chart (letters read method).
* At least a 3 month documented history of dry eye in both eyes.
* TBUT and Ocular Surface Disease Index (OSDI) Questionnaire score as specified in protocol.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Any evidence of ocular infection or inflammation within 30 days prior to Screening.
* Any ocular surgery.
* Ocular trauma requiring medical or pharmacological treatment within 1 year of Screening.
* Current presence of punctal plugs (permanent or temporary) or previous permanent punctal closure by cautery/diathermy.
* Use of topical ocular prescription or non-prescription medications within 30 days of Screening.
* Participation in any other clinical trial within 30 days prior to Screening.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lindsey, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 study centers located in the US.
Pre-assignment Details: Of the 75 enrolled, 13 participants failed to meet inclusion/exclusion criteria and were exited as screen failures prior to randomization. This reporting group includes all enrolled and randomized participants (62).
Period: Overall Study
Arm/Group | FID 119515A | Blink
Started | 43 | 19
Completed | 43 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 119515A | Blink | Total
Number analyzed (Participants) | 43 | 19 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.86) | 60.4 (14.48) | 56.4 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Tear Break-up Time (TBUT) at 60 Minutes
Description: Fluorescein dye was instilled in the eye to assess tear break-up time. After instillation of the fluorescein, the subject was instructed to blink 3 times, then stare and not blink. The investigator measured the time from the last blink until the first black (dry) spot appeared in the precorneal tear film. Tear break-up time was assessed prior to test article instillation (baseline) and at 60 minutes. Three consecutive measurements were taken per eye at each time point, with the average of the 3 scores being the value analyzed. An increase in total score equates to improvement. One eye was chosen as the study eye and only data for the study eye were used.
Time Frame: Baseline, 60 minutes
Population: This analysis population includes all randomized participants.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | FID 119515A | Blink
Number analyzed (Participants) | 43 | 19
seconds | 1.2 (0.23) | 1.2 (0.22)

2. Secondary Outcome: Area Under Curve (AUC) of TBUT From 0 to 60 Minutes
Description: Fluorescein dye was instilled in the eye to assess tear break-up time. After instillation of the fluorescein, the subject was instructed to blink 3 times, then stare and not blink. The investigator measured the time from the last blink until the first black (dry) spot appeared in the precorneal tear film. Tear break-up time was assessed prior to test article instillation (baseline) and at 5, 15, 30, and 60 minutes. Three consecutive measurements were taken per eye at each time point, with the average of the 3 scores being the value analyzed. An increase in total score equates to improvement. One eye was chosen as the study eye and only data for the study eye were used.
Time Frame: 0 to 60 minutes
Population: This analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: seconds x hours
Arm/Group | FID 119515A | Blink
Number analyzed (Participants) | 43 | 19
seconds x hours | 4.5 (0.22) | 4.5 (0.21)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (1 month). AEs were obtained through solicited and spontaneous comments from the study subjects, and through observations by the study Investigator as outlined in the study protocol.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study medication, regardless of whether or not the event had a causal relationship with the medication. This analysis group includes all subjects who received study treatment.
Arm/Group | FID 119515A | Blink
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/19
Other Adverse Events (participants affected / at risk) | 0/43 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.